CLINICAL TRIAL: NCT05617248
Title: Feasibility and Efficacy of a Brief Digital Self-efficacy Training in University Students With Self-reported Elevated Stress: A Randomized Controlled Trial
Brief Title: Feasibility and Efficacy of a Brief Digital Self-efficacy Training
Acronym: SEAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SEAPPUZH
Record Dates: First submitted 2022-09-12; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Stress; Self Efficacy
Keywords: self-efficacy, stress, digital, intervention

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial testing a brief digital intervention (SeApp) against a control group receiving only EMA
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors are blind to individuals' reports of perceived stress prior to and following the intervention, i.e. at all assessment times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Self-efficacy training (App) (Experimental): This group will receive a digital one week self-efficacy training with three training sessions per day and EMA (10 per day).
  Interventions: Behavioral: Self-efficacy App
- Control (No Intervention): This group will receive EMA questionnaires for one week (10 per day).

INTERVENTIONS:
Behavioral: Self-efficacy App — The training starts with a psychoeducational video and instructions to define two autobiographical self-efficacy The individuals will then receive three self-efficacy trainings per day based on their autobiographical memories and combined with a slow breathing exercise. Additionally, they will receive 10 daily EMA questionnaires on mood, social contacts, and virtual context.
  Arms: Experimental: Self-efficacy training (App)

SUMMARY:
The study investigates the effects of a digital, scalable self-efficacy training of repeated recall of self-efficacy memories on mental health outcomes, such as self-efficacy, anxiety, stress, hopelessness, and other mental health outcomes. A total of 94 students with elevated stress levels (≤ 13 on the Perceived Stress Scale) will be recruited and randomly assigned to training and control group. Individuals will either engage in the self-efficacy training app combined with Ecological Momentary Assessment (EMA) for 1 week (training group) or in EMA only for 1 week (control group). Baseline and post assessments will measure changes in self-efficacy, anxiety, stress, hopelessness, and other mental health outcomes.

DETAILED DESCRIPTION:
Self-efficacy is associated with positive mental health outcomes and has been proposed as a putative contributor to therapeutic outcomes in the treatment of mental health problems. It can be enhanced through experimental inductions and the recall of autobiographical mastery experiences, which have mostly been conducted in person and in the laboratory until today.

The study will investigate effects of a digital, scalable self-efficacy training of repeated recall of self-efficacy memories on mental health outcomes, such as self-efficacy, anxiety, stress, hopelessness, and other mental health outcomes. The study will recruit 94 students with elevated stress levels (≤ 13 on the Perceived Stress Scale) and randomly assigned them to training and control group. Individuals will either engage in the self-efficacy training app combined with Ecological Momentary Assessment (EMA) for 1 week (training group) or in EMA only for 1 week (control group). Baseline and post assessments will measure changes in self-efficacy, anxiety, stress, hopelessness, and other mental health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* being enrolled at a Swiss university
* aged between 18 and 29 years
* experiencing at least moderate stress (score of ≥13 on the Perceived Stress Scale
* owning a smartphone
* speaking fluent German

Exclusion Criteria:

-current psychiatric disorder

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
General self-efficacy | change from baseline to 1 day post intervention; time frame: 1 week
  The General Self-Efficacy Scale (Schwarzer & Jerusalem, 1995; Tipton & Worthington, 1984) will measure the general self-efficacy.

SECONDARY OUTCOMES:
Perceived stress | change from screening to 1 day post intervention; time frame: 1 week
  The Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983; Klein et al., 2016) will measure perceived stress.
Positive and negative affect | The Positive and Negative Affect Scale (Krohne, Egloff, Kohlmann, & Tausch, 1996; Watson, Clark, & Tellegen, 1988) will measure positive and negative affect.
  change from baseline to 1 day post intervention; time frame: 1 week
Hope | change from baseline to 1 day post intervention; time frame: 1 week
  The Trait Hope Scale (Krause, 2002; Snyder et al., 1991) will measure hope.
Depression | The Beck Depression Inventory-II (Beck, Steer, Ball, & Ranieri, 1996; Kuhner, Burger, Keller, & Hautzinger, 2007) will measure depression.
  change from baseline to 1 day post intervention; time frame: 1 week
Anxiety | change from baseline to 1 day post intervention; time frame: 1 week
  State-Trait Anxiety Inventory (Laux, Glanzmann, Schaffner, & Spielberger, 1981; Spielberger, Gorsuch, Lushene, Gagg, & Jacobs, 1983) will measure state and trait anxiety.
Hopelessness | change from baseline to 1 day post intervention; time frame: 1 week
  The Beck Hopelessness Scale (Beck, Weissman, Lester, & Trexler, 1974; Kliem, Lohmann, Mossle, & Brahler, 2018) will measure hopelessness.

OTHER OUTCOMES:
Positive and negative affect | Daily measured; changes in the course of the study participation
  EMA will capture positive and negative mood at 10 time points per day during the one week study participation. We will measure positive mood using three items (cheerful, happy, and relaxed) and negative mood using seven items (irritated, anxious, insecure, lonely, sad, overthinking, and stressed).
Dissatisfaction with social contacts | daily measured; changes in the course of the study participation
  EMA will capture dissatisfaction with social contacts at 10 time points per day during the one week study participation. There will be two options indicating dissatisfaction with social contacts: (a) being with nobody and feeling excluded or wanting to be with someone or (b) being with someone and rather wanting to be alone. We combined these into one variable.
Specific self-efficacy | daily measured in training group only; changes in the course of the study participation
  Specific self-efficacy will be captured once per day. Questions will focus on e. g. the participant's level of agreement with statements such as "Right now, I think I will be able to do what is necessary to make this training successful".
Virtual context | daily measured; changes in the course of the study participation
  EMA will capture virtual context at 10 time points per day during the one week study participation. Questions will be about who the person is with and how they feel about it.

CONTACTS AND LOCATIONS:
Locations (1):
- Birgit Kleim, Zurich, Select..., Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
It is planned to make the anonymised data available on a public repository.

REFERENCES:
- [Derived] Rohde J, Marciniak MA, Henninger M, Homan S, Ries A, Paersch C, Friedman O, Brown AD, Kleim B. Effects of a digital self-efficacy training in stressed university students: A randomized controlled trial. PLoS One. 2024 Oct 31;19(10):e0305103. doi: 10.1371/journal.pone.0305103. eCollection 2024. PMID 39480821
- [Derived] Rohde J, Marciniak MA, Henninger M, Homan S, Paersch C, Egger ST, Seifritz E, Brown AD, Kleim B. Investigating Relationships Among Self-Efficacy, Mood, and Anxiety Using Digital Technologies: Randomized Controlled Trial. JMIR Form Res. 2023 Aug 14;7:e45749. doi: 10.2196/45749. PMID 37578827